CLINICAL TRIAL: NCT01388868
Title: Determination of ED50 and ED95 of Vecuronium Infusion Dose for Maintaining Response of Train of Four Less Than 2 During the MEP Monitoring for Neurosurgery
Brief Title: Strategy for Maintaining Partial Neuromuscular Blocking Adequate for Motor Evoked Potential During Neurosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Jin Lee, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2011-04-010
Record Dates: First submitted 2011-06-28; First posted 2011-07-07 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Brain Surgery With Motor Evoked Potential Monitoring; Spine Surgery With Motor Evoked Potential Monitoring
Keywords: infusion dose; vecuronium; motor evoked potential; neuromuscular blocking agent

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TOF count guided group (Active Comparator): adjustment of neuromuscular blocking agent infusion dose every 15 minute as guided by No. of response to TOF stimulation
  Interventions: Other: TOF count guided adjustment
- T1/T0 guided group (Experimental): adjustment of neuromuscular blocking agent infusion dose every 15 minute as guided by T1 twitch height as compared with control (T0)
  Interventions: Other: T1/ T0 guided adjustment
- T2/ T0 guided group (Experimental): adjustment of neuromuscular blocking agent infusion dose every 15 minute as guided by T2 twitch height as compared with baseline (T0)
  Interventions: Other: T2/ T0 guided adjustment

INTERVENTIONS:
Other: TOF count guided adjustment — adjustment of vecuronium infusion dose every 15 minutes as guided by No. of response to TOF stimulation displayed by NMT module.
  Arms: TOF count guided group
Other: T1/ T0 guided adjustment — adjustment of vecuronium infusion dose every 15 minutes as guided by T1 twitch height as compared with baseline (T0) displayed by NMT module.
  Arms: T1/T0 guided group
Other: T2/ T0 guided adjustment — adjustment of vecuronium infusion dose every 15 minutes as guided by T2 twitch height as compared with baseline (T0)displayed by NMT module.
  Arms: T2/ T0 guided group

SUMMARY:
The maintenance of partial neuromuscular blocking during general anesthesia for neurosurgery is essential for intraoperative motor-evoked potential monitoring. However, the precise strategy of administering neuromuscular blocking agent for obtaining that goal has not been established. Therefore, the investigators tried to find the optimal initial dose of vecuronium infusion and determine the adequate goal of neuromuscular blocking as guided by neuromuscular transmission module (M-NMT Module, Datex-Ohmeda Inc, Helsinki, Finland).

DETAILED DESCRIPTION:
The maintenance of partial neuromuscular blocking during general anesthesia for neurosurgery is essential for intraoperative motor-evoked potential monitoring. However, the precise strategy of administering neuromuscular blocking agent for obtaining that goal has not been established. Therefore, the investigators tried to find the optimal initial dose of vecuronium infusion and determine the adequate goal of neuromuscular blocking as guided by neuromuscular transmission module (M-NMT Module, Datex-Ohmeda Inc, Helsinki, Finland). Previously, one to two counts of response to TOF stimulation has been considered to be primary goal of partial neuromuscular blocking needed for intraoperative motor evoked potential monitoring. However, the visualization of twitch height of response to TOF stimulation has been possible with the help of NMT module. For adequate motor evoked potential monitoring, twitch height of T1 or T2 is also as important as simple count of TOF stimulation. The investigators tried to establish a vecuronium infusion strategy as guided by not only count of TOF stimulation but also twitch height of T1 or T2.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients undergoing neurosurgery with intraoperative motor evoked potential monitoring

Exclusion Criteria:

* Patients who can not undergo motor evoked potential monitoring due to central or peripheral neuromuscular disease (e.g. Cerebral palsy, Myasthenia gravis, Acute spinal injury, neurologic shock)
* Patients with hepatic or renal disease with altered metabolism of vecuronium
* Patients with medication which influence the metabolism of vecuronium (e.g. calcium channel blocker, aminoglycoside antibiotics, Lithium, MgSO4)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Amplitude of MEP monitoring | every 30 min during MEP monitoring
  the value of MEP amplitude every 30 min during MEP monitoring

SECONDARY OUTCOMES:
latency of MEP monitoring | every 30 min during MEP monitoring
  latency of MEP monitoring every 30 min during MEP monitoring
Incidence of patient's spontaneous movement | from start to end of the MEP monitoring, an expected average of 4 hours
  Incidence of patient's spontaneous movement during MEP monitoring
Overall assessment of MEP monitoring quality | from start to end of the MEP monitoring, an expected average of 4 hours
  overall assessment of MEP monitoing quality provided by the electrophysiologist Grade I : no problem all through the monitoring Grade II : difficulty of monitoring for less than 5 min Grade III : difficulty of monitoring for 5 min to 30 min Grade IV : Difficulty of monitoring for more than 30 min
Incidence of patient's spontaneous respiration | from start to end of the MEP monitoring, an expected average of 4 hours
  Incidence of patient's spontaneous respiration as determined by end-tidal CO2 curve monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Jin Lee, M.D.,Ph.D., Principal Investigator — Samsung Medical Center; Won Ho Kim, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Jeong Jin Lee, Seoul, South Korea